CLINICAL TRIAL: NCT02958813
Title: An Integrated HIV Prevention Model for African American Mothers and Daughters
Acronym: IMARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Rush University (Other)
Responsible Party: Principal Investigator, Geri Donenberg, Associate Dean of Research, School of Public Health Professor, Department of Medicine Director, Community Outreach Intervention Projects and Healthy Youths Program, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-01627
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMARA (Experimental): IMARA blends three programs with the most relevance for AA women (SISTA) and girls (SiHLE) and families in psychiatric care (Project STYLE). Separate mother and daughter groups cover parallel content and run simultaneously, and joint activities enhance mothers' credibility as a resource for HIV/STI prevention, practice new communication skills, negotiate conflict, and strengthen the mother-daughter relationship. Activities reinforce the reciprocal impact of mothers and daughters, and enhance safe sex knowledge, attitudes, and skills. Woven throughout IMARA is the impact of alcohol and drug use on risk behavior, including condom use while high.
  Interventions: Behavioral: IMARA
- FUEL (Placebo Comparator): FUEL Health Promotion Control combines two programs, FUEL and Project Balance Health Promotion. FUEL™ promotes healthy activities by encouraging good nutrition, exercise, and informed consumer behavior. FUEL™ does not explicitly address HIV/STI prevention. Investigators will present information from Balance's session about HIV/AIDS, condoms, and other STIs. Investigators will also insert the following sessions from Balance into FUEL: alcohol use, drug/marijuana use, nutrition, exercise, and violence to increase program length.
  Interventions: Behavioral: FUEL

INTERVENTIONS:
Behavioral: IMARA — Morning and afternoon sessions begin with an icebreaker and/or poem to enhance ethnic and gender pride. IMARA's goals and motto are presented to emphasize strong mother-daughter relationships, foster sisterhood, build group cohesion, and increase motivation. Ground rules are reviewed, and each woman and girl signs the IMARA pact to confirm her commitment to the program. At the end of day 1, mothers and daughters receive homework for the week. Woven throughout IMARA is the impact of alcohol and drug use on risk behavior, including condom use while high.
  Arms: IMARA
Behavioral: FUEL — FUEL™ Health Promotion Control Group: mothers and daughters randomly assigned to FUEL™ will participate in separate 2-day workshops identical in length and intensity to IMARA. FUEL™ promotes healthy activities by encouraging good nutrition, exercise, and informed consumer behavior. Investigators will also insert the following sessions from Balance into FUEL: alcohol use, drug/marijuana use, nutrition, exercise, and violence to increase program length.
  Arms: FUEL

SUMMARY:
This study has three specific aims:

1. To conduct a 2-arm randomized controlled trial comparing IMARA to a family-based health program (FUELTM). The investigators will:

   a. Randomly assign 300 14-18 year-old AA or black girls and their primary female caregivers to IMARA (N=150) or FUELTM (N=150). Women and girls will be recruited four ways: 1) from mental health clinics using clinic liaisons, 2) flyers will be posted in clinic recruitment sites and other agencies instructing interested families to call our recruiter, 3) IMARA participants will hand flyers to interested women and girls they know, and 4) COIP field station staff will pass out flyers and recruit interested women and girls at the field stations and in the community. Investigators will examine the effects of IMARA on women and girls' sexual behavior at 6- and 12-months.
2. To evaluate the impact of IMARA on theoretical mediators posited by the Theory of Gender and Power and the Social-Personal framework associated with AA women and girls' risky sex. Investigators will:

   1. Assess changes in women and girls' Individual Attributes (HIV/AIDS knowledge, attitudes, and beliefs, mental health/emotion regulation, ethnic identity); Peer and Partner Processes (partner characteristics, relationship power dynamics, peer influences, partner communication); and Family Context (mother-daughter relationship and communication, parental monitoring) at baseline and follow-ups.
   2. Evaluate mediation and moderation of theoretical mechanisms on women and girls' sexual behavior.
3. To assess the impact of IMARA compared to FUELTM on sexually transmitted infections (STIs). Investigators will:

   1. Test women and girls' urine for three common STIs at baseline and 12-month follow up.
   2. Explore linkages between biological outcomes and targeted mediators and moderators of change.

DETAILED DESCRIPTION:
Disproportionate rates of mental illness and HIV/STIs among African Americans (AA) reflect significant health disparities. AAs account for more HIV/AIDS cases, people living with HIV/AIDS, and HIV-related deaths than any other racial group in the US. In 2004, HIV was the 3rd leading cause of death among Black women, and in 2006, AA women accounted for 66% of new AIDS cases among women. AA youth ages 13 - 19 comprise approximately 16% of US teens but 69% of new AIDS cases. Most infections among AA women and girls occur through sexual activity, and AA girls report more risky sex, less condom use, and lower perceived HIV risk than AA boys. Racial disparities also exist for AAs in rates of gonorrhea, chlamydia, and syphilis. Among 15 - 19 year old AA girls, gonorrhea rates are higher than any other race/age/gender group, and almost half of AA women have an STI. Important linkages exist between HIV/STIs and mental health; Mental illness is linked to HIV through greater risk taking, poor health promotion, and reduced effects of behavioral interventions for teens and adults.

HIV-risk factors extend beyond individual women or girls, yet few family-based, gender-specific, Afrocentric programs simultaneously address AA women, AA girls, mental health, and the mother-daughter dyad, thereby missing a critical opportunity to address HIV in a broader social context. Interventions that are sensitive to gender and culture focus on women (SISTA) or girls (SiHLE) and lack a mental health and family component. Family-based HIV prevention programs rarely address gender and culture or the adult family member's HIV risks (Project STYLE). Simultaneously targeting multiple levels in an integrated program -- the mother-daughter dyad, women, and girls -- capitalizes on the reciprocal impact of mothers and daughters, and facilitates mutual reinforcement of prevention attitudes and behavior, thereby reducing intervention decay and sustaining positive outcomes over time.

IMARA (Informed, Motivated, Aware, and Responsible about AIDS) blends gender and ethnic components of SISTA and SiHLE (gender roles, ethnic pride, relationship power) with family and mental health components from Project STYLE (affect management, parental monitoring, adolescent development, parent-child communication) to create a culturally relevant, multi-level, integrated, family-based, HIV and mental health prevention program that simultaneously targets AA women and their daughters. Based on the Theory of Gender and Power, the Social-Personal model of HIV-risk, and findings from the investigator's research, IMARA emphasizes the interplay of family, peer, partner, and individual mechanisms as mediators of sexual risk taking for women and girls. Pilot testing (N=22 dyads) revealed strong feasibility, acceptability, and tolerability: >95% consent/assent rates, 96% retention at 2-month follow-up, and very positive feedback. Promising outcome data for mothers and daughters in targeted mediators (e.g., positive attitudes about HIV/AIDS, greater intentions to use condoms, increased parental monitoring, more open mother-daughter communication, more relationship power) and sexual risk outcomes (e.g., increased condom use, fewer partners) justify a randomized controlled trial.

This study has three specific aims:

1. To conduct a 2-arm randomized controlled trial comparing IMARA to a family-based health program (FUELTM). Investigators will:

   a. Randomly assign 300 14-18 year-old AA or black girls and their primary female caregivers to IMARA (N=150) or FUELTM (N=150). Women and girls will be recruited four ways: 1) from mental health clinics using clinic liaisons, 2) flyers will be posted in clinic recruitment sites and other agencies instructing interested families to call the study recruiter, 3) IMARA participants will hand flyers to interested women and girls they know, and 4) COIP field station staff will pass out flyers and recruit interested women and girls at the field stations and in the community. Investigators will examine the effects of IMARA on women and girls' sexual behavior at 6- and 12-months.
2. To evaluate the impact of IMARA on theoretical mediators posited by the Theory of Gender and Power and the Social-Personal framework associated with AA women and girls' risky sex. Investigators will:

   1. Assess changes in women and girls' Individual Attributes (HIV/AIDS knowledge, attitudes, and beliefs, mental health/emotion regulation, ethnic identity); Peer and Partner Processes (partner characteristics, relationship power dynamics, peer influences, partner communication); and Family Context (mother-daughter relationship and communication, parental monitoring) at baseline and follow-ups.
   2. Evaluate mediation and moderation of theoretical mechanisms on women and girls' sexual behavior.
3. To assess the impact of IMARA compared to FUELTM on sexually transmitted infections (STIs). Investigators will:

   1. Test women and girls' urine for three common STIs at baseline and 12-month follow up.
   2. Explore linkages between biological outcomes and targeted mediators and moderators of change.

Hypotheses

IMARA participants will report less risky sex (fewer partners, more consistent condom use, and later sexual debut among non-sexually active girls) at 6- and 12-months and have fewer incident STI infections at 12-months; and (b) IMARA participants will report positive changes in theoretical mediators: individual attributes (more positive condom attitudes, self-efficacy, ethnic pride), peer/partner influences (more relationship power, partner communication, and awareness of partner influences on sexual decision making), mental health (improved emotion regulation and understanding of the links between mental illness and risky sex), mother-daughter communication (more open and comfortable), and mother-daughter relationships (more parental monitoring and warmth, less parental permissiveness).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls between 14-18 years of age, African American or Black.
* Women who are primary female caregivers and self-identify as African American or Black, and are over the age of 18.
* Women and daughters must agree to participate as a dyad.

Exclusion Criteria:

* If either participant is unable to understand the consent/assent process, do not speak English, are actively psychotic or severely mentally ill, or girls do not live with participating female caregiver.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Risky Sexual Behavior | From Baseline to 6 month followup
  The AIDS-Risk Behavior Assessment (ARBA) is a computer-assisted interview of sexual behavior and drug use. The ARBA was derived from five established measures used in large-scale studies to examine HIV/AIDS-risk in youth and adults. The ARBA assesses substance use, sexual behavior, and needle use. Investigators will assess mothers and daughters' condom use, sex with high-risk partners, sex while using drugs/alcohol, number of partners, sexual debut -- and relative frequency and count-based indicators.
Change in Incident STI infection | From Baseline to 12 month followup
  Investigators will measure women's and girls' STIs using biological endpoints (yes/no) to evaluate intervention effects. Investigators will screen urine for three sexually transmitted pathogens at baseline and 12- month follow up; N. gonorrhoeae, C. trachomatis, and T.vaginalis. Investigators will use nucleic acid amplification technologies (NAAT) for STI testing.
Change in Risky Sexual Behavior | From Baseline to 12 month followup
  The AIDS-Risk Behavior Assessment (ARBA) is a computer-assisted interview of sexual behavior and drug use. The ARBA was derived from five established measures used in large-scale studies to examine HIV/AIDS-risk in youth and adults. The ARBA assesses substance use, sexual behavior, and needle use. Investigators will assess mothers and daughters' condom use, sex with high-risk partners, sex while using drugs/alcohol, number of partners, sexual debut -- and relative frequency and count-based indicators.
Change in Peer and Partner Processes | From Baseline to 6 month followup
  Investigators will measure changes in women and girls' Peer and Partner Processes such as partner characteristics, relationship power dynamics, peer influences, and partner communication.
Change in Peer and Partner Processes | From Baseline to 12 month followup
  Investigators will measure changes in women and girls' Peer and Partner Processes such as partner characteristics, relationship power dynamics, peer influences, and partner communication.
Change in Individual Attributes | From Baseline to 6 month followup
  Investigators will measure changes in women and girls' Individual Attributes such as HIV/AIDS knowledge, attitudes, and beliefs, mental health/emotion regulation, and ethnic identity.
Change in Individual Attributes | From Baseline to 12 month followup
  Investigators will measure changes in women and girls' Individual Attributes such as HIV/AIDS knowledge, attitudes, and beliefs, mental health/emotion regulation, and ethnic identity.
Change in Family Context | From Baseline to 6 month followup
  Investigators will measure changes in women and girls' Individual Attributes such as Family Context (mother-daughter relationship and communication, and parental monitoring)
Change in Family Context | From Baseline to 12 month followup
  Investigators will measure changes in women and girls' Individual Attributes such as Family Context (mother-daughter relationship and communication, and parental monitoring)

IPD SHARING:
Plan to Share IPD: Undecided